CLINICAL TRIAL: NCT00101764
Title: Phase I Study of Intravitreal Injections Versus Anterior Sub-Tenon Injections of Triamcinolone Acetonide Formulation for Macular Edema in Retinal Disorders
Brief Title: Intravitreal v. Sub-tenon Injections of Triamcinolone Acetonide for Macular Edema in Retinal Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050071; 05-EI-0071
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-05-20

CONDITIONS: Macular Degeneration; Retinal Vein Occlusion; Diabetic Retinopathy
Keywords: AMD; CRVO; BRVO; Uveitis; Choroidal Neovascularization; Age-Related Macular Degeneration (AMD); Macular Edema; Central Retinal Vein Occlusion; Branch Retinal Vein Occlusion; Inflammation; Age Related Macular Degeneration; Retinal Disorder
MeSH Terms: conditions — Macular Degeneration; Retinal Vein Occlusion; Diabetic Retinopathy; Uveitis; Choroidal Neovascularization; Macular Edema; Inflammation; Retinal Diseases | interventions — Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide

SUMMARY:
The use of intravitreal injections of corticosteroid (triamcinolone acetonide) appears to be a promising treatment for a variety of ocular diseases associated with inflammation. To date, the only drug available, "Kenalog-40 Injection" produced by Bristol Myers Squibb, has not been formulated for intraocular use.

The purpose of this study is to evaluate the long-term safety and potential efficacy of novel intravitreal injections of a preservative-free formulation of triamcinolone acetonide (TAC-PF) at two dosage levels (4 mg and 8 mg) compared to anterior sub-tenon injections of TAC-PF at 20 mg.

The study will be a masked, randomized Phase I study that will enroll 120 participants with one of the following diseases: age-related macular degeneration (AMD), diabetic macular edema (DME), central retinal vein occlusion (CRVO), branch retinal vein occlusion (BRVO), or any other retinal disease with associated macular edema. At least 21 participants will be enrolled in the four designated disease strata: AMD, DME, CRVO, and BRVO. The remaining 36 participants may have one of these diseases or may be enrolled with another retinal disease. Within each disease strata, at least seven participants will be randomized to each dosing group. The participants will be randomly assigned to one of the three treatment groups.

The primary outcome will be an assessment of post-injection intraocular toxicity-related events during the 3-year follow-up, including cataract formation, development of glaucoma, and any adverse event preventing retreatment. The secondary outcomes will be an improvement in best-corrected visual acuity (BCVA, EVA) and decreases in retinal thickening and area of leakage, from baseline to year 1.

DETAILED DESCRIPTION:
The use of intravitreal injections of corticosteroid (triamcinolone acetonide) appears to be a promising treatment for a variety of ocular diseases associated with inflammation. To date, the only drug available, "Kenalog-40 Injection" produced by Bristol Myers Squibb, has not been formulated for intraocular use.

The purpose of this study is to evaluate the long-term safety and potential efficacy of novel intravitreal injections of a preservative-free formulation of triamcinolone acetonide (TAC-PF) at two dosage levels (4 mg and 8 mg) compared to anterior sub-tenon injections of TAC-PF at 20 mg.

The study will be a masked, randomized Phase I study that will enroll 120 participants with one of the following diseases: age-related macular degeneration (AMD), diabetic macular edema (DME), central retinal vein occlusion (CRVO), branch retinal vein occlusion (BRVO), or any other retinal disease with associated macular edema. At least 21 participants will be enrolled in the four designated disease strata: AMD, DME, CRVO, and BRVO. The remaining 36 participants may have one of these diseases or may be enrolled with another retinal disease. Within each disease strata, at least seven participants will be randomized to each dosing group. The participants will be randomly assigned to one of the three treatment groups. Depending on a participant's response, injections may be repeated at 3-month intervals. Participants will be followed until the last enrolled participant completes 3 years of follow-up.

The primary outcome will be an assessment of post-injection intraocular toxicity-related events during the 3-year follow-up, including cataract formation, development of glaucoma, and any adverse event preventing retreatment. The secondary outcomes will be an improvement in best-corrected visual acuity (BCVA) and decreases in retinal thickening and area of leakage, from baseline to year 1.

ELIGIBILITY:
* INCLUSION CRITERIA:

All Participants must:

1. Understand and sign the informed consent.
2. Be at least 18 years of age.
3. Have definite retinal thickening due to macular edema in the study eye, based on the clinical exam.
4. Have retinal thickness greater than or equal to 250 microns in the central subfield on OCT.
5. Have BCVA equal to or worse than 20/40 in the study eye.
6. Have sufficiently clear ocular media to permit good quality retinal photographs and angiography to allow assessment of macular area according to standard clinical practice.
7. Be able to comply with the study requirements.

EXCLUSION CRITERIA:

All participants must not:

* Have intraocular pressure greater than 25 or history suggesting glaucoma (e.g., history of the diagnosis of glaucoma, disc/nerve fiber layer defects suggestive of glaucoma) or glaucomatous visual field defects as documented by Goldmann or Humphrey perimetry taken within 6 months to qualification.

  2. Be allergic to fluorescein dyes.

  3. Have medical conditions that make consistent follow-up over the treatment period unlikely (e.g., stroke, severe MI, end-stage cancer, or history of chronic renal failure requiring dialysis or kidney transplant).

  4. Have blood pressure greater than 180/110.

  5. Be currently using or be likely to need systemic or ocular medications known to be toxic to the lens, retina, or optic nerve, such as:
  1. Deferoxamine
  2. Chloroquine/Hydroxychloroquine (Plaquenil)
  3. Tamoxifen
  4. Phenothiazines
  5. Ethambutol

     6. Have used experimental therapies for the present disease in the past 3 months.

     7. Have any contraindication to performing the necessary diagnostic procedures.

     8. Have a history of or current acute ocular or periocular infection (including any history of ocular herpes zoster or simplex).

     9. Have had any major intraocular surgical procedure within one month of enrollment.

     10. Have used systemic steroids in excess of an average 20 mg daily dose for the past 3 months.

     11. Have a known history of untoward complications from corticosteroid therapy, including elevated intraocular pressure in response to topical or periocular corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-01-05; Study Completion 2008-05-20

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bodker FS, Ticho BH, Feist RM, Lam TT. Intraocular dexamethasone penetration via subconjunctival or retrobulbar injections in rabbits. Ophthalmic Surg. 1993 Jul;24(7):453-7. PMID 8351091